CLINICAL TRIAL: NCT03952871
Title: Value of Cardiac Output Monitoring by Supra-sternal Doppler/Echocardiography in Intensive Care Unit
Acronym: SSdopler
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO18127
Record Dates: First submitted 2019-05-13; First posted 2019-05-16 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Shock
Keywords: Shock; Hemodynamic
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intensive care patient with hemodynamic instability: The study group is composed of intensive care patients which already need an invasive monitoring of the cardiac output because of a shock state.

SUMMARY:
The aim of this study is to evaluate the concordance between the measurement of cardiac blood flow by non-invasive supra sternal ultrasound and the measurements performed by invasive monitoring in intensive care patients already equipped with an invasive monitoring. This invasive monitoring consists of catheters used to measure the cardiac output allowing the supply of organs and is installed when there is need to monitor the blood flow in different hemodynamic reasons. The patient's care will not be modified, the study just requires a supplementary measure in an exam already perform in the standard care. The principal hypothesis is that we can show a concordance between this non-invasive measure and the standard invasive monitoring.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the concordance between the measurement of cardiac output by non-invasive supra sternal ultrasound and the measurements performed by invasive monitoring (trans pulmonary thermodilution or right heart catheterization) in intensive care patients already equipped with an invasive monitoring. Cross sectional study was performed in Reims university hospital. Patients who will be included in this study are patients who already have an invasive cardiac output monitoring such as trans pulmonary thermodilution or right heart catheterization for many reason as septic shock, cardiogenic shock or any shock state. Cardiac output will be measured by supra-sternal and transthoracic echography and by invasive monitoring (trans pulmonary thermodilution or right heart catheterization). Intra-class correlation coefficient will be calculated to assess the concordance between the measurement of cardiac blood flow by non-invasive supra sternal ultrasound and the measurements performed by invasive monitoring.

ELIGIBILITY:
Inclusion Criteria :

- patient admitted in intensive care unit at the Reims University Hospital and in whom invasive monitoring of cardiac output is already placed.

Exclusion Criteria:

- Age under 18 yo

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will be included in this study are patients who already have an invasive cardiac output monitoring such as trans pulmonary thermodilution or right heart catheterization for many reason as septic shock, cardiogenic shock or any shock state.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2019-04-24 (Actual); Study Completion 2019-04-24 (Actual)

PRIMARY OUTCOMES:
Concordance between the measurement of cardiac blood flow by non-invasive supra sternal ultrasound and the measurements performed by invasive monitoring | Day 0
  Value of cardiac blood flow measured by supra sternal ultrasound and invasive monitoring

SECONDARY OUTCOMES:
Concordance between the measurement of cardiac blood flow by non-invasive supra sternal ultrasound and the measurements performed by transthoracic echography | Day 0
  Value of cardiac blood flow measured by supra sternal ultrasound and thransthoracic echography

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France